CLINICAL TRIAL: NCT07390955
Title: A Phase 1 Clinical Trial to Evaluate the Safety, Pharmacokinetics, and in Vitro Neutralization of ePGT121v1-LS, PGDM1400LS, and VRC07-523LS Administered in Multiple Doses and Routes to Adult Participants Without HIV-1
Brief Title: A Study of Safety and Drug Levels of ePGT121v1-LS, PGDM1400LS, and VRC07-523LS in Adult Participants Without HIV-1
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 141/HPTN 105; 38950 (Other: DAIDS-ES ID)
Record Dates: First submitted 2025-12-22; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: HIV

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A: Group 1 (Experimental): ePGT121v1-LS 5 mg/kg to be administered via intravenous (IV) infusion at Week 0 and Week 24
  Interventions: Biological: ePGT121v1-LS (IV)
- Part A: Group 2 (Experimental): ePGT121v1-LS 20 mg/kg to be administered via IV infusion at Week 0 and Week 24
  Interventions: Biological: ePGT121v1-LS (IV)
- Part A: Group 3 (Experimental): ePGT121v1-LS 40 mg/kg to be administered via IV infusion at Week 0 and Week 24
  Interventions: Biological: ePGT121v1-LS (IV)
- Part A: Group 4 (Experimental): ePGT121v1-LS 5 mg/kg + PGDM1400LS 5 mg/kg + VRC07-523LS 5 mg/kg to be administered via IV infusion sequentially in this order at Week 0 and Week 24
  Interventions: Biological: ePGT121v1-LS (IV); Biological: PGDM1400LS (IV); Biological: VRC07-523LS (IV)
- Part A: Group 5 (Experimental): ePGT121v1-LS 20 mg/kg + PGDM1400LS 20 mg/kg + VRC07-523LS 20 mg/kg to be administered via IV infusion sequentially in this order at Week 0 and Week 24
  Interventions: Biological: ePGT121v1-LS (IV); Biological: PGDM1400LS (IV); Biological: VRC07-523LS (IV)
- Part A: Group 6 (Experimental): ePGT121v1-LS 40 mg/kg + PGDM1400LS 40 mg/kg + VRC07-523LS 40 mg/kg to be administered via IV infusion sequentially in this order at Week 0 and Week 24
  Interventions: Biological: ePGT121v1-LS (IV); Biological: PGDM1400LS (IV); Biological: VRC07-523LS (IV)
- Part B: Group 7 (Experimental): ePGT121v1-LS 375 mg (3 injections of 125 mg each) to be administered via subcutaneous (SC) injection at Week 0 and Week 12
  Interventions: Biological: ePGT121v1-LS (SC)
- Part B: Group 8 (Experimental): ePGT121v1-LS 125 mg + PGDM1400LS 100 mg + VRC07-523LS 100 mg to be administered via SC injection sequentially in this order at Week 0 and Week 12
  Interventions: Biological: ePGT121v1-LS (SC); Biological: PGDM1400LS (SC); Biological: VRC07-523LS (SC)

INTERVENTIONS:
Biological: ePGT121v1-LS (IV) — Intravenous infusion (IV)
  Arms: Part A: Group 1; Part A: Group 2; Part A: Group 3; Part A: Group 4; Part A: Group 5; Part A: Group 6
Biological: PGDM1400LS (IV) — IV infusion
  Arms: Part A: Group 4; Part A: Group 5; Part A: Group 6
Biological: VRC07-523LS (IV) — IV infusion
  Arms: Part A: Group 4; Part A: Group 5; Part A: Group 6
Biological: ePGT121v1-LS (SC) — Subcutaneous (SC) injection
  Arms: Part B: Group 7; Part B: Group 8
Biological: PGDM1400LS (SC) — SC injection
  Arms: Part B: Group 8
Biological: VRC07-523LS (SC) — SC injection
  Arms: Part B: Group 8

SUMMARY:
This study is testing a lab-made antibody called ePGT121v1-LS that targets a specific part of HIV. Researchers will give it by vein (IV) and under the skin (SC), both on its own and together with two other antibodies, VRC07-523LS and PGDM1400LS, which target different parts of the virus. They will assess safety and side effects, determine the right dose, study how the body processes the drug (pharmacokinetics or PK), and measure how well it neutralizes HIV in the blood (serum neutralizing activity). The expectation is that ePGT121v1-LS, whether given alone or with PGDM1400LS and VRC07-523LS, by IV or SC, will be safe in generally healthy adults and that the antibodies will not interfere with each other when used together.

Approximately 83 volunteers in overall good health and without HIV-1 will be enrolled into two parts (A and B).

Part A has six groups. In Groups 1-3, participants will get ePGT121v1-LS given by IV at one of three dose levels: 5 mg/kg, 20 mg/kg, or 40 mg/kg. In Groups 4-6, participants will receive three antibodies-first ePGT121v1-LS, then PGDM1400LS and VRC07-523LS-given by IV at two separate visits that are 24 weeks apart. The total study duration for participants in Part A is 48 weeks of scheduled clinic visits.

Part B has two groups. In Group 7, people will get ePGT121v1-LS as SC shots at two visits 12 weeks apart. Each visit will give a total of 375 mg, split into three injections of 125 mg each. In Group 8, people will also have two visits 12 weeks apart and will receive three antibodies as SC shots in this order: first ePGT121v1-LS (125 mg), then PGDM1400LS (100 mg), and then VRC07-523LS (100 mg). The total study duration for participants in Part B is 24 weeks of scheduled clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 55 years.
2. Can visit a participating clinic and is willing to stay in the study for its full duration.
3. Understands the study and is able and willing to give informed consent.
4. Agrees not to join another experimental study until the final required clinic visit.
5. In good overall health based on medical history, physical exam, and screening lab tests.
6. Willing to receive HIV test results.
7. Willing to discuss personal risk of getting HIV and to have HIV prevention counseling.
8. Judged by clinic staff to have a low risk of getting HIV and agrees to avoid higher risk behaviors through the last clinic visit.
9. Hemoglobin levels:

   * Women: at least 11.0 g/dL
   * Men: at least 13.0 g/dL
10. White blood cell count between 2,500 and 12,000 cells/mm³.
11. White blood cell differential is normal or acceptable to clinic staff.
12. Platelet count between 125,000 and 550,000 cells/mm³.
13. ALT (liver enzyme) less than 1.25 times the lab's upper limit of normal.
14. Creatinine (kidney test) less than 1.1 times the lab's upper limit of normal.
15. Negative tests for HIV 1 and HIV 2.
16. Negative hepatitis B surface antigen.
17. Negative hepatitis C antibody, or a negative HCV PCR if the antibody test is positive.
18. Urine protein is negative or only trace.
19. If a woman who could become pregnant: negative pregnancy test within 72 hours before the first study treatment. Women with a documented total hysterectomy, both ovaries removed, both fallopian tubes removed, or menopause (no periods for at least 1 year) do not need pregnancy testing.
20. Women who could become pregnant agree to use effective birth control for sex that could lead to pregnancy starting at least 21 days before enrollment and continuing through the last study visit.
21. Women who could become pregnant also agree not to try to become pregnant using methods like egg retrieval, artificial insemination, or in vitro fertilization starting at least 21 days before enrollment and continuing through the last clinic visit.

Exclusion Criteria:

1. Received blood products within 120 days before the first study dose (unless the safety review team approves earlier enrollment).
2. Took any experimental (investigational) research drug within 30 days before the first study dose.
3. Weighs less than 35 kg or more than 115 kg.
4. Plans to join another study using an experimental product, or any study that requires non Network HIV antibody testing, during this study.
5. Pregnant or breastfeeding.
6. Previously received an HIV vaccine in a vaccine trial. If a potential participant received placebo/control only, eligibility will be decided case by case by the safety review team.
7. Received any non HIV vaccine within 14 days before enrollment or plan to get one within 14 days after enrollment. Exception: ACAM2000 smallpox vaccine within 28 days before enrollment (or scab still present if earlier) or planned within 14 days after enrollment.
8. Received humanized or human monoclonal antibodies (mAbs), whether approved or experimental.
9. Previously received monoclonal antibodies that target HIV.
10. Receiving allergy shots within 30 days before the first study dose or scheduled within 14 days after the first dose.
11. Took immune suppressing medicines within 30 days before the first study dose. Not excluded: nasal steroid sprays; inhaled steroids (see asthma item); topical steroids for mild skin conditions; or one short course of oral/IV prednisone (less than 20 mg/day for under 14 days) finished at least 7 days before the first infusion/injection.
12. History of serious reactions to components of the study products, including anaphylaxis or symptoms like hives, trouble breathing, swelling (angioedema), or abdominal pain.
13. Received immunoglobulin within 60 days before the first study dose (separate from mAbs listed above).
14. Autoimmune disease that is not mild, stable, and uncomplicated. Mild, stable cases not needing immune suppressing drugs may be allowed if the investigator judges low risk.
15. Immunodeficiency.
16. Any significant medical issue, abnormal exam or lab result, or past condition that could:

    * Affect the immune system or its response,
    * Require medicines that affect the immune system,
    * Make repeated injections, infusions, or blood draws unsafe or not feasible (for example, very difficult veins),
    * Need active medical care to prevent serious harm during the study,
    * Have symptoms that could be mistaken for reactions to the study product,
    * Or is otherwise listed among these exclusions.
17. Any medical or skin condition, social situation, or job duty that, in the investigator's judgment, would interfere with following the study, safety assessments, or giving informed consent.
18. A psychiatric condition that prevents following the study. Specifically excluded: psychosis, current suicide risk, or a suicide attempt within the past 3 years.
19. Currently on tuberculosis treatment.
20. Asthma that is more than mild and well controlled.
21. Diabetes (type 1 or type 2). Not excluded: type 2 controlled with diet only, or a past history of gestational diabetes.
22. High blood pressure (hypertension).
23. Diagnosed bleeding disorder.
24. Cancer. Not excluded: surgically removed cancers with good assurance of cure or very low risk of recurrence during the study period.
25. Seizure disorder with any seizure in the past 3 years, or use of seizure prevention or seizure treatment medicines at any time in the past 3 years.
26. Asplenia (no functioning spleen).
27. History of widespread hives, swelling (angioedema), or anaphylaxis. Not excluded if due to a known trigger and there have been no reactions for at least 5 years, showing successful avoidance of the trigger.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of participants with solicited local Adverse Events (AEs) | Baseline through Week 48
Part B: Number of participants with solicited local Adverse Events (AEs) | Baseline through Week 24
Part A: Percentage of participants with solicited local Adverse Events (AEs) | Baseline through Week 48
Part B: Percentage of participants with solicited local Adverse Events (AEs) | Baseline through Week 24
Part A: Number of participants with solicited systemic AEs | Baseline through Week 48
Part B: Number of participants with solicited systemic AEs | Baseline through Week 24
Part A: Percentage of participants with solicited systemic AEs | Baseline through Week 48
Part B: Percentage of participants with solicited systemic AEs | Baseline through Week 24
Part A: Percentage of participants with safety laboratory abnormalities meeting grade 1 AE criteria or above | Baseline through Week 48
Part B: Percentage of participants with safety laboratory abnormalities meeting grade 1 AE criteria or above | Baseline through Week 24
Part A: Number of participants with unsolicited AEs | Baseline through Week 48
Part B: Number of participants with unsolicited AEs | Baseline through Week 24
Part A: Percentage of participants with unsolicited AEs | Baseline through Week 48
Part B: Percentage of participants with unsolicited AEs | Baseline through Week 24
Part A: Number of participants with Serious Adverse Events (SAEs) | Baseline through Week 48
Part B: Number of participants with Serious Adverse Events (SAEs) | Baseline through Week 24
Part A: Percentage of participants with Serious Adverse Events (SAEs) | Baseline through Week 48
Part B: Percentage of participants with Serious Adverse Events (SAEs) | Baseline through Week 24
Part A: Number of participants who discontinue study product administration | Baseline through Week 48
Part B: Number of participants who discontinue study product administration | Baseline through Week 24
Part A: Percentage of participants who discontinue study product administration | Baseline through Week 48
Part B: Percentage of participants who discontinue study product administration | Baseline through Week 24
Part A: Number of participants who terminate the study early | Baseline through Week 48
Part B: Number of participants who terminate the study early | Baseline through Week 24
Part A: Percentage of participants who terminate the study early | Baseline through Week 48
Part B: Percentage of participants who terminate the study early | Baseline through Week 24
Part A: Serum Concentration of ePGT121v1-LS | Baseline through Week 48
  Measured by anti-idiotype binding antibody multiplex assay
Part B: Serum Concentration of ePGT121v1-LS | Baseline through Week 24
  Measured by anti-idiotype binding antibody multiplex assay
Part A: Serum Concentration of PGDM1400LS | Baseline through Week 48
  Measured by anti-idiotype binding antibody multiplex assay
Part B: Serum Concentration of PGDM1400LS | Baseline through Week 24
  Measured by anti-idiotype binding antibody multiplex assay
Part A: Serum Concentration of VRC07-523LS | Baseline through Week 48
  Measured by anti-idiotype binding antibody multiplex assay
Part B: Serum Concentration of VRC07-523LS | Baseline through Week 24
  Measured by anti-idiotype binding antibody multiplex assay
Part A: Area Under the Concentration-Time Curve (AUC) of ePGT121v1-LS | Baseline through Week 48
Part B: AUC of ePGT121v1-LS | Baseline through Week 24
Part A: AUC of PGDM1400LS | Baseline through Week 48
Part B: AUC of PGDM1400LS | Baseline through Week 24
Part A: AUC of VRC07-523LS | Baseline through Week 48
Part B: AUC of VRC07-523LS | Baseline through Week 24
Part A: Maximum Observed Concentration (Cmax) of ePGT121v1-LS | Baseline through Week 48
Part B: Cmax of ePGT121v1-LS | Baseline through Week 24
Part A: Cmax of PGDM1400LS | Baseline through Week 48
Part B: Cmax of PGDM1400LS | Baseline through Week 24
Part A: Cmax of VRC07-523LS | Baseline through Week 48
Part B: Cmax of VRC07-523LS | Baseline through Week 24
Part A: Time to Maximum Concentration (Tmax) of ePGT121v1-LS | Baseline through Week 48
Part B: Tmax of ePGT121v1-LS | Baseline through Week 24
Part A: Tmax of PGDM1400LS | Baseline through Week 48
Part B: Tmax of PGDM1400LS | Baseline through Week 24
Part A: Tmax of VRC07-523LS | Baseline through Week 48
Part B: Tmax of VRC07-523LS | Baseline through Week 24
Part A: Clearance (CL) of ePGT121v1-LS | Baseline through Week 48
Part B: CL of ePGT121v1-LS | Baseline through Week 24
Part A: CL of PGDM1400LS | Baseline through Week 48
Part B: CL of PGDM1400LS | Baseline through Week 24
Part A: CL of VRC07-523LS | Baseline through Week 48
Part B: CL of VRC07-523LS | Baseline through Week 24
Part A: Volume of Distribution (Vd) of ePGT121v1-LS | Baseline through Week 48
Part B: Vd of ePGT121v1-LS | Baseline through Week 24
Part A: Vd of PGDM1400LS | Baseline through Week 48
Part B: Vd of PGDM1400LS | Baseline through Week 24
Part A: Vd of VRC07-523LS | Baseline through Week 48
Part B: Vd of VRC07-523LS | Baseline through Week 24
Part A: Terminal Elimination Rate Constant (λz) of ePGT121v1-LS | Baseline through Week 48
Part B: λz of ePGT121v1-LS | Baseline through Week 24
Part A: λz of PGDM1400LS | Baseline through Week 48
Part B: λz of PGDM1400LS | Baseline through Week 24
Part A: λz of VRC07-523LS | Baseline through Week 48
Part B: λz of VRC07-523LS | Baseline through Week 24
Part A: Terminal Half-life (T1/2) of ePGT121v1-LS | Baseline through Week 48
Part B: T1/2 of ePGT121v1-LS | Baseline through Week 24
Part A: T1/2 of PGDM1400LS | Baseline through Week 48
Part B: T1/2 of PGDM1400LS | Baseline through Week 24
Part A: T1/2 of VRC07-523LS | Baseline through Week 48
Part B: T1/2 of VRC07-523LS | Baseline through Week 24
Part A: Area Under the Magnitude-Breadth Curve (AUC-MB) | Baseline through Week 48
  The AUC-MB to a global panel of pseudoviruses (78) will be computed for each evaluable participant
Part B: AUC-MB | Baseline through Week 24
  The AUC-MB to a global panel of pseudoviruses (78) will be computed for each evaluable participant

SECONDARY OUTCOMES:
Serum Concentration of ePGT121v1-LS | Baseline through Week 48
  Measured by anti-idiotype binding antibody multiplex assay for all participants in all groups regardless of how many product administrations and how much product they received
Serum Concentration of PGDM1400LS | Baseline through Week 48
  Measured by anti-idiotype binding antibody multiplex assay for all participants in all groups regardless of how many product administrations and how much product they received
Serum Concentration of VRC07-523LS | Baseline through Week 48
  Measured by anti-idiotype binding antibody multiplex assay for all participants in all groups regardless of how many product administrations and how much product they received
Correlation Between Serum/Plasma Concentration and Serum Neutralization Titer (ID50) for Each Virus | Baseline through Week 48
  All participants in all groups regardless of how many product administrations and how much product they received
Correlation Between Serum/Plasma Concentration and Serum Neutralization Titer (ID80) for Each Virus | Baseline through Week 48
  All participants in all groups regardless of how many product administrations and how much product they received
Correlation Between Serum/Plasma Concentration and AUC-MB of Serum Neutralization Across the Virus Panel | Baseline through Week 48
  All participants in all groups regardless of how many product administrations and how much product they received
Area Under the Magnitude-Breadth Curve (AUC-MB) | Baseline through Week 48
  All participants in all groups regardless of how many product administrations and how much product they received
Population pharmacokinetic (PopPK) modeling of monoclonal antibody (mAb) concentration-time data | Baseline through Week 48

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Alabama CRS (Site ID: 31788), Birmingham, Alabama
  - Bridge HIV CRS (Site ID: 30305), San Francisco, California
  - The Ponce de Leon Center CRS (Site ID: 5802), Atlanta, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS) (Site ID: 30007), Boston, Massachusetts
  - Penn Prevention CRS (Site ID: 30310), Philadelphia, Pennsylvania
  - Vanderbilt Vaccine (VV) CRS (Site ID: 30352), Nashville, Tennessee
- Peru (2):
  - Via Libre CRS (Site ID: 31909), Lima Cercado, Lima region
  - Centro de Investigaciones Tecnológicas, Biomédicas y Medioambientales CRS (CITBM) - Unidad de Ensayos Clínicos (UNIDEC) (Site ID: 31970), Bellavista, Provincia Constitucional del Callao

IPD SHARING:
Plan to Share IPD: No